CLINICAL TRIAL: NCT00147095
Title: Regulation of Inflammatory Mediators in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Gene Logic (Industry)
Responsible Party: Sponsor
Other Study IDs: 02-207; DHTAB PN1259
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: COPD; Emphysema
Keywords: macrophages; neutrophils; lymphocytes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA was isolated and sent to GeneLogic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HEALTHY NON-SMOKER: Healthy non-smoker participants
- HEALTHY SMOKER: Healthy smoker participants
- COPD and smoking: Smoking participants with COPD

SUMMARY:
The aim of this study is to investigate the mechanisms whereby lung function is decreased in COPD. The hypothesis is that in diseases such as COPD, inflammatory cells including neutrophils, macrophages and lymphocytes migrate to the lung and release either more or different types of inflammatory mediators and/or destructive enzymes compared to subjects without COPD. We aim to investigate these separate cell types in the blood of subjects with COPD and identify which genes are more highly expressed when compared to cells obtained from patients without COPD. We will also investigate the lung macrophages from these subjects to identify whether the same or different genes are expressed in these cells. We will isolate different leukocyte populations from the blood and extract ribonucleic acid (RNA) from these samples. The type and quantity of RNA in these samples is a reflection of the specific genes expressed in these cells. This RNA will be sent to Gene Logic and this company will test these samples to identify which genes have been expressed. Similar experiments will be performed using macrophages obtained following bronchoalveolar lavage of these subjects. We would aim to examine the responses of leukocytes from three groups of subjects, namely (i) non-smoking controls (ii) smokers without clinical or histological signs of COPD and (iii) smokers with COPD. The isolated leukocytes will either be immediately solubilized in solutions to purify RNA or we will then use these isolated cells in vitro and following stimulation investigate whether different genes are expressed or at a differential rate in the disease state. The objective is to identify which genes are specifically expressed in patients with COPD with a view to identify novel targets for drug therapy. We will examine both leukocytes derived from peripheral blood and macrophages obtained from bronchoalveolar lavage with the aim to determine whether differences attributable to disease can be identified in both circulating cells and those at the site of disease. This is a preliminary study to determine the profile of inflammatory mediator expression from leukocytes and as such power calculations to determine the number of subjects is not appropriate.

DETAILED DESCRIPTION:
This study involves a comparison of the inflammatory responses of leukocytes derived from 3 separate subject groups. The aim of the study is to compare the responses of leukocytes from patients with COPD with subjects that smoke and healthy non-smokers. One part of the study will involve isolation of different leukocyte populations from blood from each of the subject groups. In a second part of the study, we will examine the expression of inflammatory mediators in leukocytes derived from bronchoalveolar lavage samples from patients with COPD, smokers without COPD and healthy non-smokers. In subjects that are willing to participate, we will compare blood derived leukocytes and cells derived from those undergoing BAL, although not every subject will provide both blood and BAL samples. The isolated leukocytes (both from blood and BAL) will be used for in vitro experiments to determine the differences in gene expression in inflammatory cells from patients with COPD.

Details of interventions to subjects

1. Medical History and Physical Examination A full medical history and physical examination (including height and weight) will be performed on the initial screening visit, in addition to that recorded in the clinical case notes.
2. Respiratory Assessments Forced Expiratory Volume per second (FEVI) will be measured using a dry wedge spirometer (Vitalograph, Buckingham, UK) and expressed as a percent of predicted value. Subjects will be trained in the use of the apparatus before beginning the study. The baseline value at each visit will be measured after at least fifteen minutes of quiet rest, and will be taken as the highest of three readings made at one-minute intervals. Single readings only will be taken at other times.
3. Endoscopic Bronchoscopy An operator approved by the Royal Brompton Ethics Committee will perform all bronchoscopies. The bronchoscopist that will perform these procedures is Dr Borja Cosio. Subjects will attend the bronchoscopy suite at 8.30 am after having fasted from midnight. Subjects will have pre-treatment with atropine (0.6 mg iv) and midazolam (5-10 mg iv). Oxygen (3 l/min) will be administered via nasal prongs throughout the procedure and oxygen saturation monitored with a digital oximeter. Using local anaesthesia with lidocaine (4%) to the upper airways and larynx, a fibreoptic bronchoscope (Olympus BF10 Key-Med) will be passed through the nasal passages into the trachea. Bronchoalveolar lavage (BAL) will be performed from the right middle lobe using warmed 0.9% NaCl with 4 successive aliquots of 60 ml. This is well-tolerated in subjects with COPD. Patients may experience pharyngeal irritation following the procedure; there is a 5% chance of fever following the procedure. Subjects undergoing bronchoscopy for clinical reasons will also be included in this study.
4. Venous Blood Sampling 60 ml of blood will be taken by venopuncture.

ELIGIBILITY:
Inclusion Criteria:

Healthy non-smoking subjects

All normal volunteers will meet the following criteria:

* Age 21-70 years.
* No history of respiratory or allergic disease.
* Normal baseline spirometry as predicted for age, sex and height.
* Non-smokers.
* No history of upper respiratory tract infection in the preceding six weeks.
* Not taking regular medication

COPD subjects COPD is diagnosed according to American Thoracic Society, European Respiratory Society and British Thoracic Society guidelines by the doctors in Professor Barnes' COPD clinic.

All COPD volunteers will meet the following criteria:

* Age between 40-75 years.
* A smoking history of at least 20 pack years. ( 1 pack year = 20 cigarettes per day for 1 year)
* FEV1:FVC ratio of <0.7, post-bronchodilator FEV1 of <85% predicted, reversibility with inhaled beta2-agonist of <15% of predicted FEV1: all three criteria are required.
* Current smokers or smokers who had ceased smoking for at least 6 months.
* No history of exacerbation, oral steroid or antibiotic use within the preceding 6 weeks.
* Normal serum alpha-1 antitrypsin level.
* No history of other respiratory or allergic disease.
* No evidence of atopy on skin prick testing to common aeroallergens (grass pollen, cat hair, house dust mite or Aspergillus fumigatus These tests will have already been performed as part of routine assessment in Professor Barnes' COPD clinic and we will not need to repeat them for this study.

Healthy Smokers

All healthy smoking volunteers in trials will meet the following criteria:

* Age 21-70 years.
* Smoking history of at least 10 pack years. (1 pack year = 20 cigarettes per day for 1 year).
* No history of respiratory or allergic disease.
* Normal baseline spirometry as predicted for age, sex and height.
* No history of upper respiratory tract infection in the preceding six weeks.
* Not taking regular medication.

Exclusion Criteria:

* Subjects will not included in this study if they meet any of the following exclusion criteria:
* Clinically significant findings in the medical history or on physical examination other than those of COPD in the COPD group.
* Pregnant women or mothers who are breastfeeding.
* Subjects who are unable to give informed consent.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy non-smoking and smoking subjects, smoking participants with COPD
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise E Donnelly, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital/NHLI Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No